CLINICAL TRIAL: NCT03855059
Title: Double Blind Prospective Study of IV Steroids Versus Steroids Included in Block for Orthopedic Lower Limb Surgery
Brief Title: IV Steroids Versus Steroids Included in Block for Orthopedic Lower Limb Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Peter R. Lichtenthal, MD, Professor, Anesthesiology, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 02182019
Record Dates: First submitted 2019-02-25; First posted 2019-02-26 (Actual); Results first posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Lower Limb Injury
MeSH Terms: conditions — Leg Injuries | interventions — dexamethasone 21-phosphate

STUDY DESIGN:
Intervention Model Description: Double blind study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The research pharmacist will randomize and prepare the necessary syringes for injection to look similar and have the same amount of solution as so the PI and anyone else does not know what is being given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebos (Placebo Comparator): Depending on the randomization, this group will receive a saline solution either in the IV catheter or the saline solution will be given perineural with the Mepivicaine nerve block solution.
  Interventions: Drug: Placebos
- Dexamethasone Sodium Phosphate (Active Comparator): Depending on the randomization, this group will receive dexamethasone 0.1 - 0.15 mg/kg, either in the IV catheter or the dexamethasone, 0.1 - 0.15 mg/kg will be given perineural with the Mepivicaine nerve block solution.
  Interventions: Drug: Dexamethasone Sodium Phosphate

INTERVENTIONS:
Drug: Placebos — This will be a saline solution of given IV or perineural.
  Other Names: Non-active
  Arms: Placebos
Drug: Dexamethasone Sodium Phosphate — This will be the active drug solution given IV or perineural.
  Other Names: Active treatment
  Arms: Dexamethasone Sodium Phosphate

SUMMARY:
IV and included steroids have produced the same length of block prolongation in adults as if the steroid was given with the nerve block. Clinically, this has not be noticed in children. The objective of this study is to examine this in young patients. The investigator will blindly give the steroid either in the IV or in the block solution (perineural). This is a prospective double blind study.

DETAILED DESCRIPTION:
The subject has a 50/50 chance of receiving either cohort. After the subject is randomized to receive either steroid given IV or with the nerve block, the subject is anesthetized and the subject will receive either an IV injection of 5 cc steroids or placebo, and 20 cc local anesthetic plus placebo or steroid in the nerve block, the block will be placed under ultrasound to insure proper placement of block, the dose of steroid is based on weight, 0.1 - 0.15 mg/kg. The investigator will record the time of block and IV injection. The subjects will be called by the study PI after 24 hours to determine the time of duration and again at 48 hours if needed. This is a randomized, double blind study, neither the subject or the anesthesiologist giving the injection will know what is being given. The medications will be prepared and dispensed by the Research pharmacist, a randomization chart will be obtained by the research pharmacist.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to have a lower limb Orthopedic surgical procedure.
* Scheduled to have a nerve block placed for post operative analgesia.
* American Society of Anesthesiologist (ASA) Class I - III.

Exclusion Criteria:

* Not scheduled to have a nerve block placed for post operative analgesia.

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Lichtenthal, MD, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervenous Steroid: Steroid given intervenously at the time of Peripheral nerve block
- Perineural Steroid: Steroid given in syringe with the local anesthetic
Period: Overall Study
Arm/Group | Intervenous Steroid | Perineural Steroid
Started | 25 | 25
Completed | 23 | 25
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervenous Steroid | Perineural Steroid | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Customized [Median (Full Range); unit: years]
  Population age | 13.24 [6 to 18] | 11.28 [7 to 20] | 12.26 [6 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 12 | 15 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Analgesia Duration
Description: The investigator would like to investigate if the dexamethasone given IV or with the nerve block in young patients undergoing lower limb surgery produces the same duration of analgesia.
Time Frame: 24 - 48 hours
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Intervenous Steroid | Perineural Steroid
Number analyzed (Participants) | 23 | 25
Hours | 22.1 (8.9) | 25.7 (9.8)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Followed acutely for seven days post operative and 6 months for any post op complications
Arm/Group | Intervenous Steroid | Perineural Steroid
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT03855059/Prot_SAP_000.pdf